CLINICAL TRIAL: NCT01143077
Title: A Randomized, 6-week, Open-Label, Study Evaluating The Safety, Tolerability, and Efficacy of Lurasidone for The Treatment of Schizophrenia or Schizoaffective Disorder in Subjects Switched From Other Antipsychotic Agents
Brief Title: A Study Evaluating Lurasidone for The Treatment of Schizophrenia or Schizoaffective Disorder in Subjects Switched From Other Antipsychotic Agents
Acronym: SWITCHCore
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1050289
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Lurasidone; Schizophrenia; Latuda
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lurasidone Open-Label Arm A (Experimental)
  Interventions: Drug: Lurasidone HCl
- Lurasidone Open-Label Arm B (Experimental)
  Interventions: Drug: Lurasidone HCl
- Lurasidone Open-Label Arm C (Experimental)
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — Lurasidone tablets, 40 mg/daily, 80 mg/daily, 120 mg/daily for 6 weeks
  Other Names: Latuda

SUMMARY:
Lurasidone (lurasidone HCl) is a novel psychotropic agent that is being developed as a potential new antipsychotic treatment for patients with schizophrenia. Switching between antipsychotic medications is common in the treatment of schizophrenia. The current study is designed to evaluate the effectiveness, safety, and tolerability of switching clinically stable, but symptomatic outpatients with schizophrenia or schizoaffective disorder from their preswitch antipsychotic medication to lurasidone, over a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject ≥ 18 years of age.
* Subject meets DSM-IV criteria for a primary diagnosis of schizophrenia or schizoaffective disorder.
* Subject must be judged by the investigator to be an appropriate candidate for switching current antipsychotic medication due to insufficient efficacy and/or safety or tolerability concerns.

Exclusion Criteria:

* Presence of an Axis I or Axis II disorder other than schizophrenia or schizoaffective disorder that is the primary focus of treatment prior to screening.
* Subject has experienced persistent lack of improvement in psychotic symptoms despite adequate trials (at least 6 weeks at standard doses), of two or more antipsychotic agents in the 12 months prior to screening.
* Subject is considered by the investigator to be at imminent risk of suicide or harm to self, others, or property. Subject has suicidal ideation at baseline or has attempted suicide within 90 days prior to randomization (even without hospitalization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lurasidone Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (27):
- United States (27):
  - K and S Professional Research Services, Little Rock, Arkansas
  - Synergy Clinical Research of Escondido, Escondido, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Pacific Research Partners, LLC, Oakland, California
  - California Clinical Trials, Paramount, California
  - Pasadena Research Institute, Pasadena, California
  - California Neuropsychopharmacology Clinical Research Institute (CNRI), LLC, Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Institute (CNRI), San Diego, California
  - University of California San Diego Medical Center, San Diego, California
  - Collaborative Neuroscience Network, South Bay, Torrance, California
  - Western Affiliated Research Institute, Denver, Colorado
  - Comprehensive NeuroScience, Inc., Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - Saint Charles Psychiatric Associates/Midwest Research Group, Saint Charles, Missouri
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - The Zucker Hillside Hospital, Glen Oaks, New York
  - Duke University Dept. of Psychiatry, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - CRI Worldwide - Kirkbride Center, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Wharton Research Center, Houston, Texas
  - University of Utah Hospitals and Clinics, Salt Lake City, Utah

REFERENCES:
- [Result] McEvoy JP, Citrome L, Hernandez D, Cucchiaro J, Hsu J, Pikalov A, Loebel A. Effectiveness of lurasidone in patients with schizophrenia or schizoaffective disorder switched from other antipsychotics: a randomized, 6-week, open-label study. J Clin Psychiatry. 2013 Feb;74(2):170-9. doi: 10.4088/JCP.12m07992. PMID 23473350
- [Derived] Awad G, Hassan M, Loebel A, Hsu J, Pikalov A, Rajagopalan K. Health-related quality of life among patients treated with lurasidone: results from a switch trial in patients with schizophrenia. BMC Psychiatry. 2014 Feb 23;14:53. doi: 10.1186/1471-244X-14-53. PMID 24559217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FPI June 24, 2010-LPV May 19, 2011, locations were private health clinics, university hospitals, private research facilities.
Groups:
- Lurasidone Open-Label Arm 40/40: Lurasidone 40 mg orally once daily for 14 days followed by 4 weeks of flexible dosing 40-120mg
- Lurasidone Open-Label Arm 40/80: Lurasidone 40mg for 7 days, followed by Lurasidone 80 mg for 7 days, orally once daily, followed by 4 weeks of flexible dosing 40-120mg once daily
- Lurasidone Open-Label Arm 80/80: Lurasidone 80 mg once daily orally for two weeks, followed by Lurasidone 40-120mg once daily for 4 weeks
Period: Overall Study
Arm/Group | Lurasidone Open-Label Arm 40/40 | Lurasidone Open-Label Arm 40/80 | Lurasidone Open-Label Arm 80/80
Started | 74 | 88 | 82
Completed | 58 | 73 | 67
Not Completed | 16 | 15 | 15
Not completed — Lack of Efficacy | 0 | 2 | 1
Not completed — Adverse Event | 5 | 6 | 5
Not completed — Lost to Follow-up | 2 | 3 | 4
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 3 | 3
Not completed — Non-compliance with study drug | 0 | 1 | 1
Not completed — Administrative | 1 | 0 | 0
Not completed — Principal Investigator Decision | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone Open-Label Arm 40/40 | Lurasidone Open-Label Arm 40/80 | Lurasidone Open-Label Arm 80/80 | Total
Number analyzed (Participants) | 72 | 87 | 81 | 240
Age, Categorical [Count of Participants; unit: Participants] — 244 patients were randomized, 240 received study medication.
  Participants
    <=18 years | 1 | 1 | 0 | 2
    Between 18 and 65 years | 71 | 85 | 81 | 237
    >=65 years | 0 | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] — 244 patients were randomized, 240 received study medication.
  years | 43.2 (11.3) | 44.0 (11.5) | 44.4 (10.0) | 43.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants] — 244 patients were randomized, 240 received study medication.
  Participants
    Female | 25 | 37 | 22 | 84
    Male | 47 | 50 | 59 | 156
Region of Enrollment [Number; unit: participants] — 244 patients were randomized, 240 received study medication.
  participants
    United States | 72 | 87 | 81 | 240

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse of Psychotic Symptoms During 6 Weeks
Description: Relapse is defined as any occurrence of:
  * Insufficient clinical response
  * Exacerbation of underlying disease
  * Discontinuation due to an adverse event
Time Frame: 6 Weeks
Population: Intend to treat
Measure: Mean (Standard Deviation); unit: days
Groups:
- Lurasidone Open-Label Arm 40/40: Lurasidone 40 mg daily for 14 days followed by flexible dosing between 40 and 120 mg daily for 4 weeks.
- Lurasidone Open-Label Arm 40/80: Lurasidone 40 mg daily for 7 days followed by Lurasidone 80 mg daily for 7 days followed by flexible dosing between 40 and 120 mg daily for 4 weeks.
- Lurasidone Open-Label Arm 80/80: Lurasidone 80 mg daily for 14 days followed by flexible dosing between 40 and 120 mg dailly for 4 weeks.
Arm/Group | Lurasidone Open-Label Arm 40/40 | Lurasidone Open-Label Arm 40/80 | Lurasidone Open-Label Arm 80/80
Number analyzed (Participants) | 72 | 87 | 81
days | 23.8 (12.1) | 16.9 (11.6) | 17.3 (8.9)

2. Secondary Outcome: Tolerability and Safety
Description: Number of participants with Treatment Emergent Adverse Events and Serious Adverse Events
Time Frame: 6 Weeks
Measure: Number; unit: participants
Arm/Group | Lurasidone Open-Label Arm 40/40 | Lurasidone Open-Label Arm 40/80 | Lurasidone Open-Label Arm 80/80
Number analyzed (Participants) | 72 | 87 | 81
participants | 72 | 87 | 81

ADVERSE EVENTS:
Arm/Group | Lurasidone Open-Label Arm 40/40 | Lurasidone Open-Label Arm 40/80 | Lurasidone Open-Label Arm 80/80
Serious Adverse Events (participants affected / at risk) | 3/72 | 2/87 | 0/81
Other Adverse Events (participants affected / at risk) | 45/72 | 62/87 | 59/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone Open-Label Arm 40/40 (N=72) | Lurasidone Open-Label Arm 40/80 (N=87) | Lurasidone Open-Label Arm 80/80 (N=81)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sexually inappropriate behavior (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone Open-Label Arm 40/40 (N=72) | Lurasidone Open-Label Arm 40/80 (N=87) | Lurasidone Open-Label Arm 80/80 (N=81)
Nausea (Gastrointestinal disorders) | 10 (17) | 8 (8) | 15 (23)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (7) | 7 (10)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 9 (10) | 2 (2)
Fatigue (General disorders) | 3 (3) | 5 (5) | 2 (2)
Akathisia (Nervous system disorders) | 6 (6) | 13 (17) | 11 (13)
Headache (Nervous system disorders) | 7 (13) | 10 (10) | 6 (8)
Sedation (Nervous system disorders) | 3 (3) | 2 (2) | 5 (5)
Somnolence (Nervous system disorders) | 7 (9) | 7 (7) | 2 (3)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 6 (6) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4) | 16 (16) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.